CLINICAL TRIAL: NCT02059876
Title: A Pilot Study of Dose-dense (Biweekly) Carboplatin Plus Paclitaxel With or Without Trastuzumab as Neoadjuvant Treatment for Breast Cancer
Brief Title: Dose-dense (Biweekly) Carboplatin Plus Paclitaxel With or Without Trastuzumab as Neoadjuvant Treatment for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120608
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; dose dense; neoadjuvant treatment; pathologic complete response
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — Carboplatin; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carboplatin and paclitaxel ± trastuzumab (Experimental): dose-dense(biweekly) carboplatin and paclitaxel and or without trastuzumab as neoadjuvant treatment in early breast cancer.
  Interventions: Drug: carboplatin and paclitaxel and or without trastuzumab

INTERVENTIONS:
Drug: carboplatin and paclitaxel and or without trastuzumab — dose-dense(biweekly) carboplatin and paclitaxel and or without trastuzumab as neoadjuvant treatment in early breast cancer
  Other Names: paclitaxel (Taxol); trastuzumab (Herceptine)

SUMMARY:
The purpose of this study is to determine the efficacy and safety of dose-dense(biweekly) carboplatin and paclitaxel ± trastuzumab as neoadjuvant treatment in early breast cancer.

DETAILED DESCRIPTION:
Dose-dense regimens have been shown to improve outcome when given as adjuvant therapy to patients with breast cancer compared with their three weekly counterparts. It is unknown if dose dense neoadjuvant therapy will improve survival in resectable breast cancer. This study is to evaluate the efficacy and safety of dose-dense(biweekly) carboplatin and paclitaxel ± trastuzumab as neoadjuvant treatment in early breast cancer. The endpoint of pathologic complete response is used as a surrogate marker for survival. Safety and tolerability assessed by number of grade 4 toxicities and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast carcinoma
* Clinical stage Ⅱ-ⅢB
* Patients must have measurable disease as defined by palpable lesion with both diameters ≥2cm measurable with caliper and/or a positive mammogram or ultrasound with at least one dimension ≥2cm. Bilateral mammogram and clip placement is required for study entry. Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements must have been made within the 14 days if palpable. If not palpable, a mammogram or MRI must be done within 14 days. If palpable, a mammogram or MRI must be done within 2 months prior to study entry. If clinically indicated, xrays and scans must be done within 28 days of study entry.
* Eastern Cooperative Oncology Group(ECOG) performance status 0 to 1 within 14 days of study entry
* Normal (greater than 50%) left ventricular ejection fraction (LVEF) by echocardiography
* Signed informed consent
* Adequate organ function within 2 weeks of study entry:

  1. Absolute neutrophil count >1500/mm3, Hgb >9.0 g/dl and platelet count >100,000/mm3
  2. Total bilirubin < upper limit of normal
  3. Creatinine < 1.5 mg/dL or calculated cranial cruciate ligament (CrCL) >50mL/min using the Cockcroft Gault equation
  4. serum glutamate oxaloacetate transaminase(SGOT)(AST) or serum glutamic oxaloacetic transaminase(SGPT)(ALT) and Alkaline Phosphatase must be within the range allowing for eligibility
* Patients must be over 18 years old.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Metastatic disease
* Prior chemotherapy, hormonal therapy, biologic therapy, investigational agent, targeted therapy or radiation therapy for current breast cancer. Patients with history of breast cancer greater than 5 years from initial diagnosis are eligible for the study. Patients may not have received anthracycline-based chemotherapy in the past. Patients with history of ductal carcinoma in situ(DCIS) are eligible if there were treated with surgery alone.
* History of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain disease free for greater than five years are eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Citron ML, Berry DA, Cirrincione C, Hudis C, Winer EP, Gradishar WJ, Davidson NE, Martino S, Livingston R, Ingle JN, Perez EA, Carpenter J, Hurd D, Holland JF, Smith BL, Sartor CI, Leung EH, Abrams J, Schilsky RL, Muss HB, Norton L. Randomized trial of dose-dense versus conventionally scheduled and sequential versus concurrent combination chemotherapy as postoperative adjuvant treatment of node-positive primary breast cancer: first report of Intergroup Trial C9741/Cancer and Leukemia Group B Trial 9741. J Clin Oncol. 2003 Apr 15;21(8):1431-9. doi: 10.1200/JCO.2003.09.081. Epub 2003 Feb 13. PMID 12668651